CLINICAL TRIAL: NCT04217993
Title: Jaktinib in Intermediate-risk and High-risk Myelofibrosis and Previously Treated With Ruxolitinib
Brief Title: Jaktinib for the Treatment of Ruxolitinib Intolerance of Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK006
Record Dates: First submitted 2019-11-10; First posted 2020-01-06 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Primary Myelofibrosis (PMF); Post-polycythemia Vera Myelofibrosis(Post-PV MF); Post-essential Thrombocythemia Myelofibrosis(Post-ET MF)
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Jaktinib Hydrochloride Tablets 100mg twice a day. (Experimental): This is the dose group was given Jaktinib Hydrochloride Tablets 100mg （2 tablets）dose group for twice a day.
  Interventions: Drug: Jaktinib hydrochloride tablets
- Jaktinib Hydrochloride Tablets 150mg once a day (Experimental): This is the dose group was given Jaktinib Hydrochloride Tablets 150mg （3 tablets）dose group for once a day.
  Interventions: Drug: Jaktinib hydrochloride tablets
- Jaktinib Hydrochloride Tablets 100mg once a day (Experimental): This is the dose group was given Jaktinib Hydrochloride Tablets 100mg （2 tablets） dose group for once a day
  Interventions: Drug: Jaktinib hydrochloride tablets
- Jaktinib Hydrochloride Tablets 200mg once a day (Experimental): This is the dose group was given Jaktinib Hydrochloride Tablets 200mg （4 tablets）dose group for once a day.
  Interventions: Drug: Jaktinib hydrochloride tablets

INTERVENTIONS:
Drug: Jaktinib hydrochloride tablets — Jaktinib hydrochloride tablets 100mg twice dose group，Jaktinib hydrochloride tablets 150mg qd dose group, Jaktinib hydrochloride tablets 200mg qd dose group and Jaktinib hydrochloride tablets 100mg qd dose group
  Other Names: Jaktinib

SUMMARY:
This phase IIB, open-label, multicenter study evaluated the efficacy and safety of oral Jaktinib Hydrochloride Tablets in Intermediate-risk and High-risk Myelofibrosis and Previously Treated With Ruxolitinib. The experiment is divided into two parts: dose exploration and extended research.

DETAILED DESCRIPTION:
dose exploration: It is planned to enroll about 6 subjects. According to the baseline value of platelet count at the time of enrollment, different doses (100mg Qd or 150mg Qd or 200mg Qd or 100mg Bid) of Jaktinib Hydrochloride Tablets will be Treated. The trial is in progress Adjust the dose according to relevant laboratory indicators. When at least one subject has a spleen volume reduction of ≥35% from the baseline, the sponsor and the investigator will jointly decide whether to enter the extended study part.

Extended research: It is planned to enroll about 43 subjects, and the initial dosage of Jaktinib Hydrochloride Tablets is planned to be 100mg Bid.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including the threshold value), gender is not limited;
2. Subjects diagnosed with Primary Myelofibrosis according to World Health Organization (WHO) criteria (2016 version), or diagnosed with Post-Polycythemia Vera Myelofibrosis or Post-Essential Thrombocythemia Myelofibrosis according to International Working Group Myeloproliferative Neoplasms Research and Treatment(IWG-MRT) standard. Both Janus Kinase 2(JAK2)mutation and JAK2 wild can be enrolled；
3. According to Dynamic International Prognostic Scoring System(DIPSS) , Subjects with intermediate-risk-2 or high-risk myelofibrosis were assessed, Subjects with intermediate-risk-1 myelofibrosis with hepatosplenomegaly and no response to existing treatment and requiring treatment can also be enrolled;
4. Subjects who have received or are receiving Ruxolitinib, and：Ruxolitinib treatment time is not less than 28 days; Red blood cell transfusion is still needed during treatment with Ruxolitinib; or Ruxolitinib dose (including starting dose and adjusted dose)<20mg bid，And must meet at least one of the following：Level 3 or higher platelet count reduction or Level 3 or higher anemia or Level 3 or higher hematoma/bleeding；
5. Life expectancy > 24 weeks;
6. Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 0, 1 or 2；
7. Splenomegaly: palpation of the splenic margin to or above the subcostal at least 5cm；
8. Acceptable laboratory assessments obtained within 14 days prior to enrollment:

   * Absolute neutrophil count(ANC)>0.75 x 10^9/L, blood platelet count>100 x 10^9/L;
   * Peripheral blood blast count < 10%;
   * Aspartate transaminase (AST) and alanine transaminase (ALT)≤3 x the upper limit of the normal range (ULN); Subjects with liver function impairment due to severe extramedullary haematopoiesis or iron removal therapy within 60 days prior to screening, AST and ALT≤5 x ULN; Direct bilirubin≤2.0 x ULN;
   * Calculated creatinine clearance of≥45 mL/min；
9. Meet the requirements of the Ethics Committee, voluntarily sign an informed consent form；
10. Ability to follow research and follow-up procedures.

Exclusion Criteria:

1. Any significant clinical or laboratory abnormalities that the investigator considers to affect safety assessment, such as: a. uncontrolled diabetes (> 250 mg/dL, or 13.9>mmol/L); b. had high blood pressure and antihypertensive drug treatment under two or unable to descend to the ranges (systolic blood pressure < 160 mmHg, diastolic pressure < 100 mmHg); c. peripheral neuropathy (NCI-CTC AE v5.0 grade 2 or above), etc;
2. Subjects who had a history of congestive heart failure(NCI-CTC AE v5.0 grade 3 or above), uncontrollable or unstable angina or myocardial infarction, cerebrovascular accident or pulmonary embolism in the first 6 months;
3. Screening of Subjects who have surgery within the first 4 weeks;
4. Screening for Subjects with arrhythmia requiring treatment or QTc interval (QTcB) >480ms;
5. Screening for bacterial, viral, parasitic or fungal infections that require treatment;
6. Patients which have with a history of congenital or acquired hemorrhagic diseases;(Note:With the exception of hematoma which caused by Ruxolitinib)
7. Splenectomy Subjects or in the group carried out within three months before the spleen radiation treatment (including internal radiation and external radiation)
8. Screening HIV, HBV DNA positive or higher than the normal reference range, or HCV RNA positive for HCV antibody;
9. Women who are planning to become pregnant or who are pregnant or breast- feeding, as well as those who were unable to use effective contraceptives throughout the trial;Male patients who do not use condoms during the administration and within 2 days (approximately 5 half-lives) after the last administration;
10. Subjects who have suffered from malignant tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) in the past 5 years; Combined with other serious diseases, the researchers believe that patients' safety or compliance may be affected;
11. With other serious diseases, the researchers think that may affect patient safety or compliance;
12. Subjects who had used the Jaktinib;
13. Subjects who have participated in the clinical trials of other new drugs or medical devices within the first 1 months;
14. Subjects who used the Hematopoietic growth factors within 14 days before Into the group (granulocyte growth factors, or platelet hormone) ；
15. Subjects who cannot cooperate with or cannot perform MRI or CT scans；
16. Subjects with refractory or recurrent myelofibrosis:

    refractory of myelofibrosis:After at least 28 days of adequate administration of JAK inhibitors, the spleen palpation was less than 15% smaller than before administration.Or at least 3 months later, the spleen volume on MRI/CT decreased by <10% compared with that before the administration.

    Recurrence of myelofibrosis: after at least 3 months of taking adequate amount of JAK inhibitor, the spleen was enlarged again after shrinking compared with that before taking the drug, and compared with the minimum value during taking the drug, the spleen volume increased ≥10% on MRI/CT examination or ≥30% on spleen palpation.
17. Any treatment MF medication (eg hydroxyurea,except ruxolitinib ), any immunomodulation used within 2 weeks prior to enrollment Agent (such as thalidomide), any immunosuppressant, glucocorticoids ≥ 10 mg/day of prednisone or equivalent biological strength, or Subjects within 6 half-life of the drug, over time Prevail; Subjects who had received Ruxolitinib within 1 week prior to enrolling.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Splenic response rate at Week 24 | week 24
  Splenic response rate at Week 24 is defined as the proportion of participants achieving a ≥ 35% reduction in spleen volume at Week 24 from baseline

SECONDARY OUTCOMES:
Objective response rate | up to 24 weeks
  IWG-MRT efficacy criteria
Anemia response rate | up to 24 weeks
  Proportion of anemia response in all of anemia patients
Total symptoms score(TSS) response rate | up to 24 weeks
  TSS response is defined as the proportion of subjects who achieve a ≥ 50% reduction in TSS at the Week 24 compared to baseline
Progression-free survival | up to 24 weeks
  The time from the date of enrollment to the date on which any of the following events occurred：①Spleen volume increased by ≥25% compared to the lowest value recorded during the trial including baseline；②Death from any cause
Leukemia-free survival | up to 2 years
  The time elapsed from the date of enrollment to the date of any of the following events：①The first bone marrow smear shows the date of ≥20% of the original cells；②The first peripheral blood smear showed ≥20% of the original cells and the absolute value of the original cells was ≥1×10^9/L for at least 2 weeks；③Death from any cause。
Overall survival | up to 2 years
  Time elapsed from the date of enrollment to death from any cause
Adverse event rate | up to 28 weeks
  Vital signs, physical examination, blood routine; severity and incidence of adverse events and adverse reactions (NCI-CTCAE V4.03)
Thrombotic event rate | up to 28 weeks
  Arterial thrombosis：①Coronary heart disease；②Cerebral arterial thrombosis；③Peripheral arterial occlusive disease：Such as mesenteric artery thrombosis and extremity arterial thrombosis。Venous thrombosis：①Thrombophlebitis；②Deep vein thrombosis；③Pulmonary embolism。Microcirculatory thrombosis: ① thrombotic thrombocytopenic purpura; ② hemolytic uremic syndrome; ③ extracorporeal circulation thrombosis; ④other: such as fulminant purple epilepsy and disseminated intravascular coagulation

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, Principal Investigator — The First Affiliated Hospital of Medical School of Zhejiang University
Locations (1):
- The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share date of the trial